CLINICAL TRIAL: NCT06369376
Title: A New Electrodiagnostic Approach for Pectoral Nerve Conduction Studies
Brief Title: Electrodiagnostic Approach for Pectoral Nerve Conduction Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2022-0072
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: New Nerve Conduction Protocol for Pectoral Nerve
Keywords: pectoral nerve; nerve conduction study; electromyography; electrodiagnostic; normative data

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Diagnostic Test: New nerve conduction protocol

INTERVENTIONS:
Diagnostic Test: New nerve conduction protocol — We opted for three different recording sites, each mimicking distinct parts of the pectoral muscle, allowing for a comprehensive assessment of nerve conduction across various regions.

SUMMARY:
Anatomical studies have challenged traditional perceptions of the pectoral nerve structure, revealing a network of three branches rather than the previously accepted medial and lateral branches. This study aims to explore the implications of this updated anatomy on nerve conduction studies of the pectoral nerve and proposes a modified nerve conduction study protocol to enhance diagnostic accuracy.

A study on 25 volunteers was conducted, examining the three parts of the pectoral nerve. Electrode placement followed a detailed methodology ensuring precise data collection. The nerve conduction study was performed bilaterally, exploring latency and amplitude while addressing inter-observer variability and demographic influences.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* pregnancy
* Pectoral nerve injury in the pas
* Diabetes

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Latency | 30 min
  onset latency
Amplitude | 30 min
  amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Tina Decorte, MD, Study Director — UZ Gent
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No